CLINICAL TRIAL: NCT05400863
Title: Can Sweetened Drinks Impair Therapeutic Effects of Metformin?
Brief Title: Effect of NNS on Metformin/GDF15, Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202102435
Record Dates: First submitted 2022-04-13; First posted 2022-06-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Obesity, Adolescent; Pre Diabetes
MeSH Terms: conditions — Pediatric Obesity; Glucose Intolerance | interventions — Sugar-Sweetened Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avoid Sugary Drinks and Artificially Sweetened Drinks ( plus Metformin) (Experimental): Counseling on Beverage Intake to avoid sugary sweetened and NNS (non-nutritive sweetened) drinks plus Metformin therapy (subjects will be given 12-week Metformin (500mg BID) as standard of care therapy).
  Interventions: Behavioral: avoid sugary and NNS drinks plus start Metformin
- Avoid sugary drinks only, allowed water and drinks with NNS (plus Metformin) (Active Comparator): Counseling on Beverage Intake to avoid sugary drinks (allowed water and drinks sweetened with NNS) plus Metformin therapy (subjects will be given 12-week Metformin (500mg BID) as standard of care therapy).
  Interventions: Behavioral: avoid sugary drinks (allowed water and drinks sweetened with NNS) plus start Metformin

INTERVENTIONS:
Behavioral: avoid sugary and NNS drinks plus start Metformin — Subjects will receive education and counseling to avoid all sweetened drinks (drink water only). Participants will be asked to consume minimum of 3 drinks/day
  Arms: Avoid Sugary Drinks and Artificially Sweetened Drinks ( plus Metformin)
Behavioral: avoid sugary drinks (allowed water and drinks sweetened with NNS) plus start Metformin — Subjects will avoid drinks sweetened with sugar (can have diet drinks sweetened with NNS). Participants will be asked to consume minimum of 3 drinks/day
  Arms: Avoid sugary drinks only, allowed water and drinks with NNS (plus Metformin)

SUMMARY:
Metformin use for diabetes has the benefit of causing weight loss in some. The investigators in a preclinical trial, demonstrated that mice consuming non-nutritive sweetened (NNS) drinks had worse glucose improvements and weight loss than mice consuming sugar drinks or water. This study will conduct a pilot to determine if this translates into pediatric clinical practice. The hypothesis is that NNS drinks impair metformin-induced satiation, weight loss, and glucose tolerance.

DETAILED DESCRIPTION:
This study will enroll 40 children ages 10-21 years (will be recruited from the University of Florida (UF) Pediatric Obesity& Metabolic clinic in Gainesville) and randomize eligible participants into a 2-arm, 12-week Metformin (500mg BID) intervention (n=20/group) in which one arm will be randomized to receive education and counseling to avoid all sweetened drinks (drink water only) and the other to avoid drinks sweetened with sugar (can have diet drinks sweetened with NNS). Participants will be asked to consume minimum of 3 drinks/day In the initial visit (baseline visit) the investigators will do a complete evaluations of physical health and eating behaviors. The investigators will draw lab work including A1c and GDF15 levels. The investigators will also get anthropometric measurements of height and weight to calculate body mass index (BMI). For assessment of beverage intake, the investigators reviewed questionnaires validated in children and adolescents in the past 10 years to better reflect currently available beverages. The investigators combined data from BEVQ-15 (that was validated in children aged 6-18 years) and BFQ(17 items questionnaire validated in young adults, aged 16-30 years),and edited further to make the important distinction between unsweetened and artificially sweetened drinks while adding several examples to each category to help improve correct selection. The investigators will also limit to weekly intake assessments. Data will be collected biweekly. Following completion of the 12-week intervention, participants will return fasting to assess the effectiveness of the metformin treatment on the following: hemoglobin A1C (A1c), Growth Differentiation Factor 15 (GDF15), with BMI and 24-hour dietary recall, including questions about change in hunger while on metformin. The investigators predict that metformin-induced GDF15 levels will be blunted in participants consuming NNS beverages. To improve compliance and decrease attrition, The investigators will provide performance feedback and interpretation of physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will have already been prescribed Metformin as part of their normal clinical care
* Must also be aged 10-21 years
* Have a diagnosis of obesity (BMI > 95th%ile or >30 kg/m2 - whichever is lower) and pre-diabetes (A1c between 5.7 and 6.4%)

Exclusion Criteria:

* Previous treatment with oral hypoglycemic medications, (2) resting systolic blood pressure (SBP)>180 mm/Hg or diastolic blood pressure (DBP)>100mm/Hg, (3) self-reported pregnancy

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
change in BMI z-score between the two groups at 12 weeks | 12 weeks
  Compare post-intervention (metformin) body weight between participants randomized to receive education and counseling to either a) avoid all sweetened drinks (drink water only) or b) avoid drinks sweetened with sugar (can have diet drinks sweetened with NNS)

SECONDARY OUTCOMES:
improvement of A1C due to metformin between the 2 groups at 12 weeks | 12 weeks
  Compare post-intervention change in glycemic control between participants randomized to receive education and counseling to either a) avoid all sweetened drinks (drink water only) or b) avoid drinks sweetened with sugar (can have diet drinks sweetened with NNS)

OTHER OUTCOMES:
metformin-induced rise in GDF15 in both groups at 12 weeks | 12 weeks
  Compare post-intervention rise in GDF15 between participants randomized to receive education and counseling to either a) avoid all sweetened drinks (drink water only) or b) avoid drinks sweetened with sugar (can have diet drinks sweetened with NNS)

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Bernier, MD, Principal Investigator — University of Florida; Esraa Ismail, MD, Principal Investigator — University of Florida
Locations (1):
- UF pediatric metabolic and obesity clinic, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided